CLINICAL TRIAL: NCT07299565
Title: Analysis of Immunological and Pharmacological Aspects Regarding Infection Free Survival After Surgical Treatment of a Periprosthetic Knee Infection During Hospitalization: a Microdialysis Study
Brief Title: Analysis of Pharmacological Aspects Regarding Infection Free Survival After Surgical Treatment of a Periprosthetic Knee Infection: a Microdialysis Study
Acronym: PJI_K_MD
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Alexander Franz, Dr. med., B. Sc., University Hospital, Bonn
Other Study IDs: 2025_B_PJI_Knee
Record Dates: First submitted 2025-08-25; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-08

CONDITIONS: Periprosthetic Knee Infection
Keywords: two-stage exchange; infection; PJI; microdialysis; infection free survival; treatment monitoring; muscle mass; patient reported outcom measures; bone cement
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients presenting with an infected knee prosthesis

SUMMARY:
This study aims to use the technique of microdialysis to analyse the intraarticular space of the knee joint after removal of a periprosthetic joint infection affected endoprosthesis and implantation of an antibiotic-containing cement spacer over the entire period of the first hospitalization (usually 14 days) to closely monitor pharmacological and immunological aspects. In detail, antibiotic concentrations in the joint cavity and systemic circulation will be assessed according to reinfection rates, infection-free survival and fucntional outcome over a 12-month folluw-up period.

DETAILED DESCRIPTION:
Periprosthetic joint infection (PJI) of the knee is a severe complication following joint arthroplasty, with rising incidence and reinfection rates as high as 30-35 % despite the widely used two-stage revision approach (DOI: 10.36186/reporteprd112025). This treatment combines systemic antibiotic treatment and local therapy via antibiotic impregnated bone cement - so called spacers. During a first surgery the infected prosthesis is removed and a temporary spacer is implemented. It is either preformed for hip joints or intra operatively formed for knee joints and used to temporarily fill the joint cavity and stabilize the joint. Both spacer designs include the same antibiotics gentamicin and vancomycin. After six to eight weeks, during which systemic antibiotics (e.g. cefuroxime, cefazolin) are applied for two weeks and continued orally, the spacer is removed in a second surgery and a new prosthesis is implemented into a pathogen free compartment. With this treatment patients often experience prolonged immobility, delayed rehabilitation, and reduced quality of life, along with causing significant healthcare costs (DOI: 10.1016/j.jiph.2020.09.006, 10.3389/fmed.2021.552669,10.1016/j.joca.2017.07.022). Despite clinical relevance, there is a lack of in vivo data on sustained and therapeutic local antibiotic elution during spacer implantation and their correlation with clinical outcomes. A previous pilot study by the same research group used the technique of microdialysis for 72 hours postoperatively, only on patients with PJI of the knee (DOI: 10.3390/antibiotics14080742). It showed microdialysis as a feasible method and displayed fast declining, yet therapeutic concentrations eluted from the spacer for 72 hours. Microdialysis is a technique to continuously generate samples from interstitial fluid of human tissue based on the principle of passive diffusion along a semipermeable membrane (DOI: 10.1016/j.xphs.2016.08.016).

This study now aims to extend the surveillance period to 14 days postoperatively and investigate the intraarticular compartment knee joints during PJI treatment with two-stage revision. Microdialysis will be used again to measure locally eluted antibiotic concentrations as well as inflammatory markers. Furthermore, during the second surgery intraarticular samples will be taken intraoperatively to look at antibiotic concentrations six weeks at spacer removal. Found antibiotic concentrations will be correlated to reinfection rates at 12 months following two-stage revision. Furthermore, the quality of life and functional recovery in regard to infection-free survival and local antibiotic levels will be investigated. For this, functional testing (e.g., 6-Minute-Walking-Test, Timed-Up-And-Go) as well as patient reported outcome measures (e.g. SF-36, Knee/Hip Injury and Osteoarthritis Outcome Score) will be used and information will be gathered before and at multiple follow-up time points until 12 months after surgery. By using two different spacer designs (e.g., surgeon made vs. manufacture-made) elution kinetics and concentration levels will be examined based on process of preparation.

The correlation of antibiotic findings with clinical and patient-reported outcomes seeks to fill a critical knowledge gap regarding the pharmacological efficacy of spacers in two-stage revision.

ELIGIBILITY:
Inclusion Criteria:

* clinical indication for two-stage revision of knee PJI
* approval for surgery by the orthopedic and anesthesiologic department
* being over 18 years of age
* written, informed consent after detailed patient information about the study protocol and possible study dependent risks

Exclusion Criteria:

* known allergies to antibiotics gentamicin and vancomycin used within the spacer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 30 patients over 18 years of age presenting with PJI after total knee arthroplasty and indication for prosthesis explantation and temporary spacer implantation
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-11-15 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Intraarticular concentrations of local antibiotics | Pre-Surgery (prothesis removal), during 14 days of hospitalization as well as pre-surgery of the reimplantation (approx. six weeks after the first surgery)
  Microdialysis will help to generate intraarticular hip joint samples after removal of an infectes prosthesis and spacer implantation. These samples will be analysed for spacer eluted antibiotics.

SECONDARY OUTCOMES:
Comparison intraarticular antibiotic concentrations to venous blood concentrations | Pre-Surgery (removal of the prothesis), during hospitalization of 14 days and before reimplantation of the prothesis.
  Antibiotic concentrations measured in intraarticular samples generated by microdialysis will be compared to venous blood serum concentrations

OTHER OUTCOMES:
Correlation between infection free survival and antibiotic concentrations | Preoperatively, during hospitalisation, preoperatively before the second surgery and at follow up time points (6 weeks, 3 months, 6 months, 12 months).
  Analyzed concentrations of local and systemic antibiotic concentrations will be correlated with infection free survival within the follow up (infection free survival: successfull wound healing, no signs of lossening within X-rays, no increase of inflammatory markers).

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Bonn, Bonn, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No